CLINICAL TRIAL: NCT04485377
Title: Assessing Californians Communities' Experiences With Safety Net Supports Survey
Brief Title: Safety Net Support Use in California
Acronym: ACCESS
Status: Completed | Type: Observational
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 048228-001
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Households
Keywords: poverty; child health; safety net programs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator's goal is to promote equity by understanding the drivers of disparities in access to income support, particularly among urban and rural Latinx, African American, and white populations in California (CA). This study aims to capture levels of awareness, barriers to uptake, and the benefits of participation in the Earned Income Tax Credit (EITC), a tax credit for low- to moderate-income working individuals and families, among households with children ages 0-5 years old. To achieve this goal, the investigators will conduct a mixed-methods, cross-sectional, descriptive study in three diverse counties in California: Los Angeles (urban, nearly half Latinx), Alameda (urban, ethnically diverse), and Merced (rural, predominantly Latinx and white).

DETAILED DESCRIPTION:
Using both focus groups and survey interviews, the investigators will recruit parents of young children (ages 0-5) eligible for the EITC (confirmed with screening questions regarding age, family size, marital status, and income) who either: 1) have utilized the program, or 2) have not utilized the program (do not file taxes or filed taxes but have not filed for EITC benefits). For the first group, the investigators will probe the value of the EITC benefits for their families, what experiences they had filing their taxes and receiving the benefit, how they spent the EITC benefits, and their thoughts about alternative approaches for benefit delivery that would better support their families. For the second group, the investigators aim to understand what they have heard of the program, why they may not have taken advantage of the benefits, and their recommendations for making the program more accessible. The investigators will also explore how EITC take-up varies by demographic variables, such as county of residence, income, and race/ethnicity, as well as children's and parents' characteristics, and enrollment in other programs designed to support low-income families with young children. The investigators will also ask questions about families' experiences with COVID-19 and related mitigation strategies (e.g. school closures, etc). As described in greater detail below, all data collection activities will be conducted in partnership with agencies such as WIC and Head Start, and through partnerships with the University of California Cooperative Extension program and other similar agencies.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children 0-6
* Lives in Alameda, Merced of Los Angeles counties
* Income below certain cut-offs

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families living with low-income, in three selected counties in California
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Poverty: survey | Baseline
  Income Assets Food insecurity (USDA 6-Item Food Security Module, range=0-6 with 0=high food security and 6=very low food security) Food resources
Employment: survey | Baseline
  Employment type and status over the past year, earned/unearned income, transfers
Safety net participation and perceptions of participation: survey | Baseline
  Safety net program participation & enrollment in programs, such as Special Supplemental for Women, Infants, and Children (WIC), Supplemental Nutrition Assistance Program (SNAP), Unemployment Insurance, Medi-Cal, Children's Health Insurance Program (CHIP), Covered CA, and paid sick leave and other poverty alleviation programs, perceived barriers, amount of benefits received, stigma (Welfare Stigma Scale: 6-item Treatment Welfare Stigma Scale, a multiple choice format questionnaire, possible scores 6-30, with 30 representing high stigma towards participating in welfare programs from other individuals.)
Mental health: survey | Baseline
  CES-D - Center for Epidemiologic Studies- Depression scale (Depression Scale: 10-item Center for Epidemiologic Studies Depression Scale (CESD-10), a multiple choice format questionnaire, possible scores 0-30, with 30 representing a high risk of depression diagnosis.
  Generalized Anxiety Disorder Scale: 7-item Generalized Anxiety Disorder Scale (GAD-7), a multiple choice format questionnaire, possible scores 0-21, with 21 representing a high risk of generalized anxiety diagnosis.
Physical Health: survey | Baseline
  Adult and child self-rated health, comparing self-rated health to 12 months ago, occurrence of health, developmental, emotional, or behavioral problem.
Health care utilization: survey | Baseline
  Health care utilization, insurance, concerns about affording healthcare, last visit with a healthcare provider, delays in receiving healthcare, forgoing healthcare.
COVID-19-related questions | Baseline
  Effect on employment and income, essential worker, childcare/schooling, shelter-in-place, housing stability and changes, experiences with racial discrimination, risk for contracting COVID-19, ability to self-isolate, ability to partake in behaviors to prevent spread of COVID-19. Questions pulled from two different surveys: The Epidemic/Pandemic Questionnaire and COVID-19 Community Outcome Surveys.
Tax Credit Question | Baseline
  Self-perceived awareness, eligibility, participation, sources of information, intended vs actual spending patterns of Federal Earned Income Tax Credit (EITC), CA EITC, Young Child Tax Credit (YCTC), and federal child tax credit (CTC), resources used to file taxes, reasons for participation or lack of participation
2018 and 2019 Tax Return Data: survey | Baseline
  Awareness of tax filing deadline changes, tax filing status, number of dependents, EITC receipt, amount of EITC received, adjusted gross income, federal CTC receipt, amount of federal CTC received CA EITC receipt, amount of CA EITC receipt, YCTC receipt, amount of YCTC received.

SECONDARY OUTCOMES:
Racial discrimination: survey | Baseline
  Perception of safety, major experiences of racial discrimination, minor experiences of racial discrimination. Questions pulled from Major Experiences of Discrimination Scale and Racial Microaggressions Scale.
Housing: survey | Baseline
  Housing status, house ownership/characteristics, current living situation, access to bathrooms, housing crowding, housing quality, cross streets, zip code, rent payment amount, frequency of rent payments, rental assistance program participation, trouble paying utilities, living in a "doubled up" arrangement, letting others live with them in a "doubled up" arrangement, history of homelessness in childhood, history of homelessness in adulthood
Attitudinal variables: survey | Baseline
  Attitudes about public assistance, civic engagement, role of government
Food insecurity: survey | Baseline
  Food Insecurity Survey: 6-item Food Insecurity Scale, a multiple choice format questionnaire, possible scores 0-6, with 6 representing very low food insecurity.
  Food Insecurity Survey - Kids Module: 9 additional questions to assess childrens' food insecurity.
  Self-perceived food insecurity comparison to 12 months ago Changes in food-related habits. Questions pulled from United Nations Standing Committee on Nutrition.
Housing-related changes from Coronavirus pandemic (COVID-19): survey | Baseline
  Ability to pay rent, application to emergency housing money, reasons for not applying to emergency funding, number of moves, reasons for moves (e.g. difficulty paying rent, eviction), knowledge of eviction moratoriums, legal assistance seeking behavior
Demographic information: survey | Baseline
  Gender, age, education level, race/ethnicity, marital status, number of children, birthplace, language spoken at home. Questions were pulled from National Health Interview Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Berkeley School of Public Health, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No